CLINICAL TRIAL: NCT00099645
Title: A Randomized, Placebo-Controlled, Phase I/II Trial of the Anti-HIV Activity and Safety of VGX-410 (Mifepristone) at Three Dose Levels in HIV-1 Infected Subjects
Brief Title: Anti-HIV Activity and Safety of 3 Different Doses of Mifepristone in HIV Infected People
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5200; 10186 (Registry Identifier: DAIDS ES); ACTG A5200
Record Dates: First submitted 2004-12-17; First posted 2004-12-20 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Mifepristone; Mifeprex; RU486; VGX-410; Abortion Pill; Investigational Drug
MeSH Terms: conditions — HIV Infections | interventions — Mifepristone

INTERVENTIONS:
Drug: Mifepristone

SUMMARY:
The purpose of this study is to determine the anti-HIV activity and safety of 3 different doses of mifepristone (also known as VGX-410 and RU486) in HIV infected people.

Hypothesis: Mifepristone will be generally safe (no serious adverse effects) and well tolerated.

DETAILED DESCRIPTION:
Mifepristone is a potent anti-glucocorticoid compound that effectively inhibits replication of both laboratory and clinical HIV isolates in vitro. This study will evaluate the anti-HIV activity and safety of 3 different doses of mifepristone in HIV infected people.

This study will last approximately 2 months. Participants will be randomly assigned to one of 4 study arms, and will receive either mifepristone or placebo daily for 28 days. Arm A participants will receive one of three doses of placebo; Arm B participants will receive 75 mg mifepristone; Arm C participants will receive 150 mg mifepristone; and Arm D participants will receive 225 mg mifepristone. A thorough neck and thyroid examination will be performed within 30 days prior to study entry. Blood collection and vital signs measurement will occur at study entry and Days 3, 7, 14, 21, 28, and 56. Urine collection and pill counts will also be done at some study visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* CD4 count of 350 cells/mm3 or more within 90 days prior to study entry
* HIV-1 viral load of 2000 copies/ml or more within 90 days prior to study entry
* Willing to use acceptable forms of contraception during the study and for 30 days after stopping study medication
* If currently taking precautionary concomitant medications, must be on stable doses for more than 8 weeks prior to study entry and have no plans to change medications or doses for the duration of the study
* Body weight at least 40 kg (88 lbs) within 90 days prior to study entry

Exclusion Criteria:

* Antiretroviral treatment (ART) within 16 weeks prior to study entry, or intend to start ART within 60 days after entry
* Adrenal disorders
* History of autoimmune endocrine disease in self or family
* History of active hepatitis B or C
* Current treatment for hepatitis B or C
* Moderate to severe liver disease
* Blood disorders or current anticoagulant therapy
* Prior pituitary tumor, surgery, radiation treatment, or pituitary failure
* Moderate to large goiters or thyroid nodules
* Diabetes mellitus
* Unusual uterine bleeding within 12 months prior to study entry
* Current hormonal contraception or intrauterine (IUD) use, including progesterone-containing vaginal rings
* Pregnancy within 90 days prior to study entry
* Breast-feeding
* Drugs that act as inhibitors or inducers of metabolism by cytochrome P450 3A4
* Systemic corticosteroids or hormonal agents within 90 days prior to study entry
* Any immunomodulator, HIV vaccine, or investigational therapy within 90 days prior to study entry
* Any vaccination within 30 days prior to study entry
* Systemic cytotoxic chemotherapy within 90 days prior to study entry
* History of allergy to mifepristone or the study formulations
* Current drug or alcohol abuse that, in the opinion of the investigator, may interfere with the study
* Any other conditions that may interfere with participant evaluation during the study
* Serious illness requiring systemic treatment or hospitalization. Patients who complete therapy or are clinically stable on therapy for at least 14 days prior to study entry are not excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Changes in HIV-1 viral load from baseline to Days 14 and 28

SECONDARY OUTCOMES:
Within 28 days on study, occurrence of toxicity, rash, and symptoms of adrenal insufficiency, including fatigue, nausea, anorexia, vomiting, and dizziness
changes from baseline viral load on Days 7, 14, 21, 28, and 56
pre-dose concentrations of mifepristone on Days 14 and 28 and serum level of alpha-1 acidic glycoprotein (AAG) at Day 0
percentage and counts of CD4 and CD8 cells at baseline and on Days 14, 28, and 56
Vpr amino acid sequences on Days 0, 14, 28, and 56
comparison of the magnitude and diversity of effector T cell response to HIV antigens at Days 0, 28, and 56
change in fasting concentrations of plasma insulin, free fatty acids, high-density lipoprotein (HDL) cholesterol and triglycerides, and in insulin sensitivity between Days 0 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Michael F. Para, MD, Study Chair — Ohio State University
Locations (10):
- United States (10):
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - Georgetown University CRS (GU CRS), Washington D.C., District of Columbia
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Washington U CRS, St Louis, Missouri
  - Unc Aids Crs, Chapel Hill, North Carolina
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - Univ. of Pennsylvania Health System, Presbyterian Med. Ctr., Philadelphia, Pennsylvania
  - Pitt CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Schafer E, Wagner M, and Ayyavoo V. Antiviral Effects of Mifepristone and its Analogs on HIV-1 Vpr-Induced Virus Replication. 11th Conference on Retroviruses and Opportunistic Infections. February 2004.
- [Background] Ayyavoo V, Mahboubi A, Mahalingam S, Ramalingam R, Kudchodkar S, Williams WV, Green DR, Weiner DB. HIV-1 Vpr suppresses immune activation and apoptosis through regulation of nuclear factor kappa B. Nat Med. 1997 Oct;3(10):1117-23. doi: 10.1038/nm1097-1117. PMID 9334723
- [Result] Para MF, Schouten J, Rosenkranz SL, Yu S, Weiner D, Tebas P, White CJ, Reeds D, Lertora J, Patterson KB, Daar ES, Cavert W, Brizz B; ACTG A5200 Team of the ACTG. Phase I/II trial of the anti-HIV activity of mifepristone in HIV-infected subjects ACTG 5200. J Acquir Immune Defic Syndr. 2010 Apr 1;53(4):491-5. doi: 10.1097/QAI.0b013e3181d142cb. PMID 20130470